CLINICAL TRIAL: NCT06508125
Title: Comparing the Efficacy of Cross-Linked and Non-Cross-Linked Hyaluronic Acid in Treating Subdeltoid Bursitis: A Double-Blind, Randomized Clinical Trial
Brief Title: Cross-linked and Non-cross-linked Hyaluronic Acid in Subdeltoid Bursitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024SKHADR036
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Subdeltoid Bursitis; Hyaluronic Acid
Keywords: Subdeltoid Bursitis; Hyaluronic acid; cross linked
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cross-linked hyaluronic acid group (Experimental): cross-linked hyaluronic acid injection, one-time, plus physical therapy
  Interventions: Drug: cross-linked hyaluronic acid
- non-cross-linked hyaluronic acid group (Active Comparator): non-cross-linked hyaluronic acid injection, one-time, plus physical therapy
  Interventions: Drug: non-cross-linked hyaluronic acid

INTERVENTIONS:
Drug: cross-linked hyaluronic acid — cross-linked hyaluronic acid injection with physical therapy
  Other Names: physical therapy
  Arms: cross-linked hyaluronic acid group
Drug: non-cross-linked hyaluronic acid — non-cross-linked hyaluronic acid injection with physical therapy
  Other Names: physical therapy
  Arms: non-cross-linked hyaluronic acid group

SUMMARY:
This study aims to compare the efficacy of different structures of hyaluronic acid, namely cross-linked and non-cross-linked hyaluronic acid, in treating subdeltoid bursitis.

DETAILED DESCRIPTION:
A double-blind, randomized clinical trial will be conducted to collect 52 patients with subdeltoid bursitis. The patients will be injected with cross-linked or non-cross-linked hyaluronic acid under ultrasound guidance. Before treatment, one week after treatment (i.e., one week after injection), one month after treatment, and three months after treatment to detect shoulder pain (visual analog scale; pressure ergometer to measure pain pressure threshold), function (including Disabilities of the Arm, Shoulder, and Hand: DASH and Shoulder Pain and Disability Index: SPADI), quality of life (Brief version of the World Health Organization Quality of Life Scale: WHOQOL-BREF) will be arranged.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of subdeltoid bursitis
* age 20 or older 20
* at least one positive in the painful arc, neer test, or Hawkins test
* can attend three months of intervention and follow-up

Exclusion Criteria:

* history of malignancy
* previous shoulder operation or injury
* previous shoulder injections in the past three months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder pain and disability, ranges from 0-100, higher scores indicate more pain or disability

SECONDARY OUTCOMES:
Disabilities of the arm, shoulder, and hand | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure sports/music and work related to shoulder pain, ranges from 0-100, higher scores indicate more pain or disability
Visual analog scale | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder pain, ranges from 0-10, higher score indicate more pain
range of motion | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder range of motion, higher score indicate higher range of motion
Brief version of the World Health Organization Quality of Life Scale | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure quality of life, ranges from 0-100, higher scores indicate better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No